

| Study title | Lessening the impact of fatigue in inflammatory rheumatic diseases: a randomised | | | | | | |
|---|---|---|---|---|---|---|---|
| Name of CI: | clinical trial (LIFT) IRAS 216267 Prof Gary J Macfarlane | | | | | | |
| | l ioi Gaily G | Madranand | | | | | |
| Participant ID: | | | | | | | |
| Please initial each box | | | | | | | Initial |
| 1. I <b>confirm</b> that I have re | | • | | | • | ). I have | |
| had the opportunity to consider the information, ask questions and have had these answered satisfactorily. I understand that I can contact the study team if I have any further questions. | | | | | | | |
| 2. I understand that my pa | articipation is v | oluntary and t | hat I am | free to | withdraw at any time, | without giving any | |
| reason, without my medical care or legal rights being affected. I agree that any information collected prior to my withdrawal will be used in the analysis; however, no new | | | | | | | |
| information will be collec | | prior to my w | itnorawa | I WIII DE | e used in the analysis; | nowever, no new | |
| 3. I agree that relevant sec | ctions of my me | edical notes a | nd data | collecte | ed during the study, ma | ay be looked at by | |
| individuals from the University of Aberdeen and collaborators involved in the study, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. | | | | | | | |
| I give permission for th | | - | | | | | |
| 4. I agree to be contacted | by the study te | am via post, t | elephon | e or en | nail after the trial perio | d is over. | |
| I <b>agree</b> that identifiable contact information will be kept after the end of this study and this information will be held confidentially and securely in accordance with the data protection act. | | | | | | | |
| held confidentially and s | securely in acco | ordance with t | he data | protect | ion act. | | |
| 5. I give permission for the LIFT study research group to contact my GP or other health care professional to | | | | | | | |
| let them know I am takir | ng part in this re | esearch. | | | | | |
| 6. I give permission for th | e LIFT study re | esearch group | to notify | mv GF | P and/or my health care | e team if incidental | |
| findings are discovered. | - | ocaron group | 10 110111 | y O. | anarer my nearm ear | y tourn in inforderital | |
| <b>5</b> | | | | | | | |
| Please initial <b>one</b> box only | of the arouns t | hat will get th | eranist. | Helivere | ed treatment. I do give | nermission to the | Initial |
| 7. If I am allocated to one of the groups that will get therapist-delivered treatment, I do give permission to the<br>LIFT trial research group to record some of the sessions (phone or internet-based audio/video calls) for<br>quality assurance purposes only. | | | | | | | |
| If I am allocated to one of the groups that will get therapist-delivered treatment, I do not give permission to | | | | | | | |
| LIFT trial research group to record any of the sessions (phone or internet-based audio/video calls). | | | | | | | |
| Please initial box | | | | | | | Initial |
| 8. I <b>agree</b> to take part in the | is randomised | study. | | | | | |
| 9. OPTIONAL - I agree that | at data collecte | d as part of th | nis study | may b | e linked to with health | research datasets | |
| and data from other rese | | | | | | | |
| Please initial <b>one</b> box only | | | | | | | Initial |
| 10. I agree to give additional blood samples for future ethically approved studies, together with the related data, | | | | | | | |
| and I <b>understand</b> it may be linked with health research datasets and data from other research studies. My unique NHS number may be used to do this. | | | | | | | |
| I <b>do no</b> t agree to give an additional blood sample for future ethically approved studies. | | | | | | | |
| 3 3 | | , | | , | | | |
| Name of participant | Dat | e (DD/MON/YY | YY) | | Signature | | |
| | | (0.0.10.10.10.10.10.10.10.10.10.10.10.10. | 200 | | | | |
| Name of person taking consent | Dat | e (DD/MON/YY | YY) | | Signature | | |

NOTE: Original for local Investigator Site File, copies for participant, for central Trial Master File and for participant's medical notes